CLINICAL TRIAL: NCT00851955
Title: Role of CXCR2 Ligands/CXCR2 Biological Axis in Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Massimo Raimondo, M.D., PI, Mayo Clinic
Other Study IDs: 07-000099
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Pancreatitis; Pancreatic Cancer
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 1. Normal pancreas patients: Patients with no documented clinical history of pancreatic diseases supported by at least 1 negative imaging test (EUS, CT scan or MRI).
- 2. Chronic pancreatitis patients: Patients with documented diagnosis of moderate to advanced chronic pancreatitis supported by at least 1 positive imaging test (EUS,CT scan or MRI).
- 3. Pancreatic cancer patients: Patients with documented tissue diagnosis (or clinical suspicion) of Pancreatic Cancer.

SUMMARY:
The investigators hypothesize that the CXCR2 ligands/CXCR2 biological axis plays an important role in promoting angiogenesis in PC; and that the genetic changes and the microenvironment of the tumor regulate the expression of CXCR2 ligands/CXCR2 in PC in order to potentiate their angiogenic phenotype. A corollary of this hypothesis is that the cell surface receptors (CXCR2) and the intracellular signaling pathways that mediate the angiogenic responses induced by ELR+ CXC-chemokines are potential targets for novel therapeutic interventions in PC.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects - No documented clinical history of pancreatic diseases supported by at least 1 negative imaging test. (EUS, Ct scan or MRI)
* Chronic pancreatitis - Documented diagnosis of moderate to advanced chronic supported bpancreatitisy at least 1 positive imaging test. (EUS, Ct scan or MRI)
* Pancreatic Cancer - Documented tissue diagnosis (or clinical suspicion) of Pancreatic Cancer.

Exclusion Criteria:

* Exclusion criteria will include age younger than 18 yrs, pregnancy, previous pancreatic or gastric resection, and inability to tolerate routine endoscopy with conscious sedation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
All cause mortality | One year

SECONDARY OUTCOMES:
For pancreatic patients from whom tissue samples will be available, we will examine the association between presence/absence of each marker in the tissue versus the marker level in blood and in pancreatic juice. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Raimondo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States